CLINICAL TRIAL: NCT06160492
Title: Phase III Clinical Trial Evaluating the Efficacy of 5-aminolevulinic Acid (5-ALA HCl) Fluorescence-guided Microsurgery Versus Conventional White Light Microsurgical Resection in Patients With Malignant Gliomas (WHO Grade 3/4)
Brief Title: Phase III Clinical Trial Evaluating the Resection Efficacy of 5-Aminolevulinic Acid Hydrochloride (5-ALA HCl) Fluorescence-Guided Microsurgery Versus Conventional White Light Microsurgery in Patients With Malignant Glioma (WHO Grade 3/4)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ALA HCl-LEES-2022-01
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: 5-aminolevulinic Acid; Fluorescence-guided Resection
MeSH Terms: interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, open, parallel-group, multicenter, conventional treatment-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- test group (Experimental): The test group was set to administer a dose of 20 mg/kg body weight, and 3 hours before anesthesia (range 2-4 hours), 5-ALA HCl was dissolved in drinking water and taken orally, after which they underwent fluorescence-guided resection of malignant gliomas
  Interventions: Drug: 5-aminolevulinic acid
- control group (No Intervention): The control group was operated by traditional white light microscope tumor resection, and all tumor tissues were removed as far as possible within the safety range. Cranial enhancement MRI was performed within 72h after surgery .

INTERVENTIONS:
Drug: 5-aminolevulinic acid — Patients were randomly assigned to 5-aminolevulinic acid (20 mg/kg bodyweight）Those randomly allocated to 5-aminolevulinic acid were scheduled to receive freshly prepared solutions of 5-aminolevulinic acid orally 3 h (range 2-4) before induction of anaesthesia. Solutions were prepared by dissolving the contents of a vial (1·5 g) in 50 mL of drinking water.
  Other Names: 5-ALA HCl
  Arms: test group

SUMMARY:
This is a randomized, open, parallel-group, multicenter clinical trial evaluating 5-aminolevulinic acid (5-ALA HCl) oral solution with powdered fluorescent microscopic tumor resection versus white light microscopic tumor resection in patients with malignant gliomas (WHO grade 3/4).

DETAILED DESCRIPTION:
As specified in the trial procedure, patients entered the screening period after signing an informed consent form, and subjects who met the inclusion criteria and did not meet the exclusion criteria were randomly divided into two groups and randomized 1:1. The test group received 5-ALA HCl administration + excision under fluorescence and the control group received excision under white light. The test group was set to administer a dose of 20 mg/kg body weight, and 3 hours before anesthesia (range 2-4 hours), 5-ALA HCl was dissolved in drinking water and taken orally, after which they underwent fluorescence-guided resection of malignant gliomas. The light source is switched by the surgeon according to the intraoperative situation. Try to remove all tumor tissues within the safe range. The first 10 subjects in the test group underwent pharmacokinetic testing. Cranial enhanced MRI was performed within 72 h after surgery.

In the control group, traditional white light microscopic tumor resection surgery was used, and pathological specimen tissues were retained according to pathological SOPs, and all tumor tissues were resected as far as possible within a safe range. Cranial enhancement MRI was performed within 72h after operation

During the course of the trial, subjects were monitored for adverse events (AEs) from 4h prior to the administration/surgery of the test drug to the end of the postoperative safety follow-up period and recorded in the EDC, all AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18-70 years of age, inclusive;
* Patients with presumably new malignant gliomas (WHO grade 3/4) diagnosed by imaging;
* have a Karnofsky Performance Status (KPS) ≥ 60;
* Ability to take oral medications;
* Laboratory tests meeting the following criteria within ≤ 7 days preoperatively:

Alanine aminotransferase (ALT), Mentholatum aminotransferase (AST), Glutamyl transpeptidase (GGT) < 100 IU/L; Serum total bilirubin (TBIL) < 51.3 μmol/L (3.0 mg/dl); Serum creatinine (CRE) < 176.8 μmol/L (2.0 mg/dl);

* Non-surgically sterilized or female subjects of childbearing potential need to have a negative serum pregnancy test result and must be non-lactating females; female subjects of childbearing potential and male subjects whose spouses are of childbearing potential are voluntarily using contraception for a period of 3 months after administration of the test drug;
* Subjects are able to understand the informed consent form, voluntarily participate and sign the informed consent form, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

* Known hypersensitivity to the test drug ingredients, aminoglutaric acid, porphyrins, or their analogs;
* acute or chronic porphyria; history of cutaneous photosensitivity, actinic dermatoses, and exfoliative dermatitis
* Tumor located in the midline, basal ganglia, cerebellum, or brainstem;
* Inability to undergo enhanced MRI (pacemaker, contrast allergy, and other reasons);
* Subjects taking other trial medications within 30 days prior to the start of this trial or subjects undergoing other clinical trials at the same time;
* Comorbid uncontrolled cardiac conditions such as: a) New York Heart Association (NYHA) class ≥II, b) severe/unstable angina, c) primary cardiomyopathy, d) myocardial infarction or previous coronary/peripheral artery bypass grafting within ≤6 months prior to the procedure, e) difficult-to-control hypertension, f) severe arrhythmia requiring medication or intervention, and g) screening echocardiographic left ventricular ejection fraction <50%;
* Active hepatitis B or C (unless HBV-DNA titers below the minimum detection limit and HCV-RNA negative on antiviral therapy can be included), HIV-positive or known history of acquired immunodeficiency syndrome;
* Any other condition that, in the opinion of the investigator, makes participation in the trial inappropriate;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
gross total resection rate(GTR rate） | Within 72 hours after surgery
  Proportion of subjects in the test and control groups whose tumors were determined to have met the criteria for complete resection by cranial enhancement MRI within 72 hours postoperatively

SECONDARY OUTCOMES:
Positive diagnostic rate of strongly fluorescent tissue biopsy specimens | Within 15 days after surgery
  Proportion of tissue specimens taken intraoperatively in the test group that were positive for tumor by pathological testing

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Province Tumor Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No